CLINICAL TRIAL: NCT01104337
Title: Dose-dependent Drug-drug Interaction Between Paracetamol and Warfarin in Adults Receiving Long-term Oral Anticoagulants: A Randomized Controlled Trial
Brief Title: Drug Interaction Between Paracetamol and Warfarin
Acronym: INPAWA2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Pr Stephane Mouly, Therapeutic Research Unit, Department of Internal Medicine, Hospital Lariboisière, Paris,France
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: INPAWA2-URT
Record Dates: First submitted 2010-04-12; First posted 2010-04-15 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-02

CONDITIONS: Deep Venous Thrombosis; Pulmonary Embolism; Atrial Fibrillation; Stroke; Antiphospholipid Syndrome
Keywords: paracetamol; warfarin; drug interaction; pathogenic mechanism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Atrial Fibrillation; Stroke; Antiphospholipid Syndrome | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paracetamol 2g/d (Experimental): 18 patients on stable warfarin therapy received a 10-day regimen of paracetamol 2g/d
  Interventions: Drug: paracetamol
- Paracetamol 3g/d (Experimental): 18 patients on stable warfarin therapy received a 10-day regimen of paracetamol 3g/d
  Interventions: Drug: paracetamol
- Placebo (Placebo Comparator): 9 patients on stable warfarin therapy received a 10-day regimen of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: paracetamol — Treatment consisted of two paracetamol 500mg (Doliprane® 500mg, Sanofi-aventis, Paris, France) tablets twice a day along with two matching placebo tablets once daily
  Arms: Paracetamol 2g/d
Drug: paracetamol — Treatment consisted of two paracetamol 500mg (Doliprane® 500mg, Sanofi-aventis, Paris, France) tablets three times a day
  Arms: Paracetamol 3g/d
Drug: Placebo — Treatment consisted of two matching placebo tablets three times a day.
  Arms: Placebo

SUMMARY:
The objective of this study is to investigate whether paracetamol, given at therapeutic doses (2g/day and 3 g/day), may potentiate the anticoagulant effect of warfarin.

DETAILED DESCRIPTION:
Paracetamol is recommended as a first-line analgesic and antipyretic therapy in patients receiving short- and long-term oral anticoagulation, especially elderly patient.However,Increased INR was previously observed in patients treated with warfarin and paracetamol given at the maximum recommended dose (4g/day).

To date, the mechanism of this interaction has not been determined.A recent in vitro study suggested that the toxic metabolite N-acetyl-para-benzoquinoneimine (NAPQI) appeared to interfere with vitamin K-dependent γ-carboxylase (VKD-carb) and vitamin K epoxide reductase (VKOR) activites12. The question remaining to be dealt with is whether this in vitro observation can explain the in vivo paracetamol-warfarin interaction. We aim to evaluate the effect of paracetamol at the most widely used doses 2 and 3g/day on INR in stable patients treated with warfarin in a double blind randomized placebo-controlled trial and to identify the mechanism involved in this interaction in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with warfarin (target INR 2 to 3) stable anticoagulation at 2 to 9 mg for more than 30 days
* Aged 18 years or older
* Laboratory values (hemoglobin, blood cell counts, albumin, blood ionogram, complementary hemostasis parameters and aspartate, alanine transaminases (AST and ALT))remained within normal limits

Exclusion Criteria:

* Any treatment change within 7 days before enrollment
* Any paracetamol intake within the last 14 days
* Drug allergy Concomitant drug ( 5-fluorouracile, acetylsalicylic acid, non steroidal anti-inflammatory drugs, chloramphenicol, diflunisal, miconazole)
* St John's wort treatment
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-03; Primary Completion 2008-11 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The mean maximum increase in INR from baseline to Day 10 (INR (max-D1)) | 10 days

SECONDARY OUTCOMES:
The mean maximum INR (INRmax) | 10 days
The time to the first variation of INR observed | 10 days
Day 10 - Day 1 differences in factors II, V, VII, AT-III plasma concentrations between groups. | 10 days
Day 10 - Day 1 differences in paracetamol plasma concentration between groups. | 10 days
Day 10 - Day 1 differences in R(-), S(-)warfarin plasma concentrations between groups. | 10 days
Day 10 - Day 1 differences in Gla-type Osteocalcin (Gla-OC) and undercarboxylated Osteocalcin (Glu-OC)plasma concentrations between groups. | 10 days
Relation between age and the mean maximum increase in INR from baseline to Day 10 (INR (max-D1) | 10 days
  Relation between age and INR (max-D1)is measured using regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Mouly, MD, PhD, Principal Investigator — Therapeutic Research Unit, Department of Internal Medicine, Hospital Lariboisière, Paris, France; Guy Simoneau, MD, Principal Investigator — Therapeutic Research Unit, Department of Internal Medicine, Hospital Lariboisière, Paris, France
Locations (1):
- Therapeutic Research Unit, Department of Internal Medicine, Hospital Lariboière, Paris, France